CLINICAL TRIAL: NCT04679766
Title: Evaluation of Ice Cream Cone Technique as a Flapless Guided Bone Regenerative Method With Immediate Implant Placement in Management of Patients With Labial Plate Dehiscence: A Case Series
Brief Title: Evaluation of Ice Cream Cone Technique With Immediate Implant Placement in Patients With Labial Plate Dehiscence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Amagad, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAmagad
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Dental Implant; Guided Bone Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with non-restorable tooth in maxillary bi-cuspid region with labial/buccal plate dehiscence (Experimental)
  Interventions: Procedure: Ice cream cone technique with immediate implant as a flapless bone regenerative method in management of patients with labial plte dehiscence

INTERVENTIONS:
Procedure: Ice cream cone technique with immediate implant as a flapless bone regenerative method in management of patients with labial plte dehiscence — Atraumatic extraction will be done The extraction socket will be debrided to remove any residual debris using surgical curettes Socket walls will be checked using a periodontal probe to ensure integrity of all sockets walls except the labial bone plate which must show a dehiscence. Implant placement will be done. All implants will engage at least 3 mm apical to the apical end of the socket with adequate primary stability Resorbable collagen membrane will be cut confirming to the size and shape of the defect of labial bone plate dehiscence. The membrane will be placed against internal surface of the extraction socket against the remaining buccal plate of bone. The gap between the collagen membrane and the implant fixture will be filled with xenograft particulates.The membrane will be folded in palatal direction to seal the socket in an ice cream cone shape, then will be secured using non-resorbable sutures

SUMMARY:
Immediate tooth replacement with immediate implants into fresh extraction sockets has become a common and promising clinical procedure in daily practice in regard of implant survival, osseointegration and esthetic outcomes . However, there are some challenges encountered in the treatment of patients with labial bone plate dehiscence. Deficiency of facial bone anatomy has a negative impact on esthetics and is a critical causative factor for esthetic implant complications and failures ..

Few studies investigated the reconstitution of labial bone plate dehiscence using ice cream cone technique and their results showed adequate bone regeneration 4 to 6 months where no labial plate was present prior to grafting technique. Ice cream cone technique as a flapless grafting technique in conjunction with immediate implant placement in patients with labial bone plate dehiscence requires further studies for its clinical relevance and approval.

DETAILED DESCRIPTION:
Classical methods of guided bone regenerative methods succeeded to partially reconstitute the lost labial plate of bone using different grafting materials with barrier membranes.

This might be attributed to the necessity of using a full mucoperiosteal flap which interrupts the vascular supply to the bone and jeopardizing the process of total facial bone regenerative process. Therefore, Tan-Chu et al., (2014) described in a case report an innovative technique using resorbable collagen membrane in the shape of ice cream cone and allograft in the reconstitution of labial plate in patients with socket type II after extraction with folding the membrane to seal the socket and containing the blood clot to allow for occupation of osteogenic cell population without raising a flap. This technique showed an adequate bone regeneration with net result of 1.32 mm prior to no labial plate present before grafting. Hence, using immediate implant placement with the conjunction of the ice cream cone technique in regeneration of labial plate of bone needs to be further assessed to evaluate its clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Non-restorable teeth in maxillary inter-bicuspid region.
2. All teeth have labial plate dehiscence (socket type II) after extraction.
3. Patients free from any systemic conditions that may affect healing.
4. Adequate bone volume for the placement of immediate implant.
5. Presence of the adjacent teeth.
6. Compliant patients.

Exclusion Criteria:

1. Smokers.
2. Pregnant females.
3. Patients who were taking or currently taking any of the bisphosphonates.
4. Any disease that might affect bone metabolism as osteoporosis.
5. Insufficient inter-occlusal distance or mesio-distal space to place an implant supported restoration.
6. The presence of any signs of acute infection in the surgical site or the adjacent natural teeth.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Changes in buccal/labial vertical bone dimensions | 6 months post operative
  Vertical bone dimension will be measured at day 0 and 6 months post-operative

SECONDARY OUTCOMES:
Changes in labial/buccal plate thickness | 6 months
  Measured at day 0 and 6 months post-operative using Cone beam tomography
Keratinized tissue width | 6 months
  Measured using william's graduated probe
Gingival thickness | 6 months
  Measured using william's graduated probe
Post operative pain measured with VAS scale | 1 week -2 weeks
  VAS scale from 0 to 10, where 0 no pain and 10 with highest pain
Post-operative patient satisfaction with Yes or No question | 6 months
  Yes or No question of overall patient satisfaction of the procedure

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, informed consent and clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study
Access Criteria: Clinicaltrials.gov
URL: http://ClinicalTrials.gov